CLINICAL TRIAL: NCT06348199
Title: A Phase III Randomised, Double-blind, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity Between SB27 (Proposed Pembrolizumab Biosimilar) and Keytruda in Subjects With Metastatic Non-squamous Non-small Cell Lung Cancer
Brief Title: A Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity Between SB27 and Keytruda in Subjects With Metastatic Non-squamous Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB27-3004
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SB27 (Experimental): SB27 will be administered followed by Pemetrexed and Carboplatin (Carboplatin will be administered for the first 4 cycles).
  Interventions: Drug: SB27
- Keytruda (Active Comparator): Keytruda will be administered followed by Pemetrexed and Carboplatin (Carboplatin will be administered for the first 4 cycles).
  Interventions: Drug: Keytruda

INTERVENTIONS:
Drug: SB27 — Will be administered intravenously at a fixed dose of 200 mg every 3 weeks
  Arms: SB27
Drug: Keytruda — Will be administered intravenously at a fixed dose of 200 mg every 3 weeks
  Arms: Keytruda

SUMMARY:
The goal of this clinical trial is to confirm that SB27 works in the same way as Keytruda in metastatic non-squamous non-small cell lung cancer (NSCLC) patients. The main question it aims to answer is:

• How effective the study drug is Participants will receive either investigational product (SB27 or Keytruda) and chemotherapy every 3 weeks.

Researchers will compare SB27 and Keytruda to see if SB27 works in the same way as Keytruda.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Have been diagnosed with stage IV non-squamous NSCLC
* Have not received any prior systemic anti-cancer therapy for metastatic NSCLC
* Agree to use adequate methods of contraception

Exclusion Criteria:

* Unable or unwilling to take folic acid and vitamin B12 supplementation
* Severe hypersensitivity to treatment with another monoclonal antibody, any ingredient contained in SB27 or Keytruda, or any component of platinum-containing compounds or pemetrexed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) at Week 24 | At Week 24
  Defined as the proportion of subjects achieving a complete response (CR) or partial response (PR) at Week 24 according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (94):
- Bosnia and Herzegovina (3):
  - SB Investigative Site, Banja Luka
  - SB Investigative Site, Mostar
  - SB Investigative Site, Sarajevo
- Brazil (9):
  - SB Investigative Site, Curitiba
  - SB Investigative Site, Florianópolis
  - SB Investigative Site, Ijuí
  - SB Investigative Site, Natal
  - SB Investigative Site, Pelotas
  - SB Investigative Site 1, Porto Alegre
  - SB Investigative Site 2, Porto Alegre
  - SB Investigative Site, Rio de Janeiro
  - SB Investigative Site, Santo André
- Georgia (7):
  - SB Investigative Site, Batumi
  - SB Investigative Site 1, Tbilisi
  - SB Investigative Site 2, Tbilisi
  - SB Investigative Site 3, Tbilisi
  - SB Investigative Site 4, Tbilisi
  - SB Investigative Site 5, Tbilisi
  - SB Investigative Site 6, Tbilisi
- Germany (4):
  - SB Investigative Site, Düsseldorf
  - SB Investigative Site, Halle
  - SB Investigative Site, Moers
  - SB Investigative Site, Neuss
- India (10):
  - SB Investigative Site, Bangalore
  - SB Investigative Site, Bhubaneshwar
  - SB Investigative Site, Bhubaneswar
  - SB Investigative Site, Erandwane
  - SB Investigative Site, Hyderabad
  - SB Investigative Site 1, Jaipur
  - SB Investigative Site 2, Jaipur
  - SB Investigative Site, Mumbai
  - SB Investigative Site, Sūrat
  - SB Investigative Site, Udaipur
- Japan (10):
  - SB Investigative Site, Himeji
  - SB Investigative Site, Iwakuni
  - SB Investigative Site, Izumi
  - SB Investigative Site, Kawachi-Nagano
  - SB Investigative Site, Kobe
  - SB Investigative Site, Kochi
  - SB Investigative Site, Sagamihara
  - SB Investigative Site, Tachikawa
  - SB Investigative Site, Takarazuka
  - SB Investigative Site, Toyonaka
- Malaysia (6):
  - SB Investigative Site, George Town
  - SB Investigative Site, Johor Bahru
  - SB Investigative Site, Kota Bharu
  - SB Investigative Site, Kuantan
  - SB Investigative Site, Lembah Pantai
  - SB Investigative Site, Putrajaya
- Mexico (3):
  - SB Investigative Site, Aguascalientes
  - SB Investigative Site, Guadalajara
  - SB Investigative Site, Mexico City
- Philippines (5):
  - SB Investigative Site, Davao City
  - SB Investigative Site, Makati City
  - SB Investigative Site, Manila
  - SB Investigative Site, Quezon City
  - SB Investigative Site, San Juan City
- Romania (8):
  - SB Investigative Site, Cluj-Napoca
  - SB Investigative Site 1, Craiova
  - SB Investigative Site 2, Craiova
  - SB Investigative Site, Craiova
  - SB Investigative Site, Iași
  - SB Investigative Site, Oradea
  - SB Investigative Site, Sibiu
  - SB Investigative Site, Suceava
- Serbia (5):
  - SB Investigative Site 1, Belgrade
  - SB Investigative Site 2, Belgrade
  - SB Investigative Site, Kamenitz
  - SB Investigative Site, Kragujevac
  - SB Investigative Site, Niš
- Spain (7):
  - SB Investigative Site, Leganés
  - SB Investigative Site, Málaga
  - SB Investigative Site, Ourense
  - SB Investigative Site, Oviedo
  - SB Investigative Site, Santiago de Compostela
  - SB Investigative Site, Seville
  - SB Investigative Site, Valencia
- Thailand (4):
  - SB Investigative Site 1, Bangkok
  - SB Investigative Site 2, Bangkok
  - SB Investigative Site, Bangkok Noi
  - SB Investigative Site, Khon Kaen
- Turkey (Türkiye) (13):
  - SB Investigative Site, Adapazarı
  - SB Investigative Site 1, Ankara
  - SB Investigative Site 2, Ankara
  - SB Investigative Site, Bağcılar
  - SB Investigative Site, Balgat
  - SB Investigative Site, Çubuk
  - SB Investigative Site, Istanbul
  - SB Investigative Site, İzmit
  - SB Investigative Site, Kavaklıdere
  - SB Investigative Site, Konak
  - SB Investigative Site, Maltepe
  - SB Investigative Site, Seyhan
  - SB Investigative Site, Sivas